CLINICAL TRIAL: NCT05203575
Title: Building a Behavioural Intervention Programme to Improve Self-Management of Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Singapore Health Services (Other)
Responsible Party: Principal Investigator, Lawrence Jin, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: DCOF
Record Dates: First submitted 2021-12-02; First posted 2022-01-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Control (No Intervention): Control condition
- Weekly nudge in Cycle 2 (Experimental): Weekly nudge intervention in Cycle 2
  Interventions: Behavioral: Goal-Setting plus Weekly Nudge in Cycle 2
- Fast-forwarding (Experimental): Fast-forwarding interventions in both Cycles
  Interventions: Behavioral: Fast-forwarding in Cycle 1; Behavioral: Fast-forwarding in Cycle 2
- Fast-forwarding with weekly nudge in Cycle 2 (Experimental): Fast-forwarding interventions in both Cycles, plus weekly nudge intervention in Cycle 2
  Interventions: Behavioral: Fast-forwarding in Cycle 1; Behavioral: Fast-forwarding in Cycle 2; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 2
- Weekly nudge in Cycle 1 (Experimental): Weekly nudge intervention in Cycle 1
  Interventions: Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1
- Weekly nudge (Experimental): Weekly nudge interventions in both Cycles
  Interventions: Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 2
- Fast-forwarding with weekly nudge in Cycle 1 (Experimental): Fast-forwarding interventions in both Cycles, plus weekly nudge intervention in Cycle 1
  Interventions: Behavioral: Fast-forwarding in Cycle 1; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1; Behavioral: Fast-forwarding in Cycle 2
- Full intervention (Experimental): All interventions applied in all Cycles
  Interventions: Behavioral: Fast-forwarding in Cycle 1; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1; Behavioral: Fast-forwarding in Cycle 2; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 2
- Fast-forwarding in Cycle 1 (Experimental): Fast-forwarding intervention in Cycle 1
  Interventions: Behavioral: Fast-forwarding in Cycle 1
- Full in Cycle 1 (Experimental): Fast-forwarding and weekly nudge interventions in Cycle 1
  Interventions: Behavioral: Fast-forwarding in Cycle 1; Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1

INTERVENTIONS:
Behavioral: Fast-forwarding in Cycle 1 — The fast-forwarding intervention will consist of a projection of future risk of co-morbidities. A visual projection model will be built using archival data available through the Singapore Diabetes Registry. The projection model will use the current profile of the participant to calculate a risk profile for the participant's potential complications and co-morbidities, which will be presented as a pie chart. The tool will also present alternative scenarios to the participant and visualize how the likelihood of complications or co-morbidities would decrease or increases if his/her habits changed. This will provide the motivational aspect of the intervention.
  This intervention takes place during Cycle 1 (first 14 weeks).
  Arms: Fast-forwarding; Fast-forwarding in Cycle 1; Fast-forwarding with weekly nudge in Cycle 1; Fast-forwarding with weekly nudge in Cycle 2; Full in Cycle 1; Full intervention
Behavioral: Goal-Setting plus Weekly Nudge in Cycle 1 — The procedure for goal-setting will start with the participant receiving a list of possible goals. The moderator will go through the list with the participant to identify which goals the participant is comfortable with and could reasonably achieve, and to tick off those goals that the participant has already achieved. The participants will choose their own goals. In each subsequent week, the moderator will check-in with the participant and tick off the goal(s) that have been achieved.
  Chat groups of 10-15 people will be formed to administer the weekly nudge. The participants will be encouraged to introduce themselves and to interact with each other during each the chat session. Every week for the following 14 weeks, the moderator will post diabetes-related content on the WhatsApp chat group and introduce topics of interest according to a planned schedule.
  This intervention takes place during Cycle 1 (first 14 weeks).
  Arms: Fast-forwarding with weekly nudge in Cycle 1; Full in Cycle 1; Full intervention; Weekly nudge; Weekly nudge in Cycle 1
Behavioral: Fast-forwarding in Cycle 2 — The fast-forwarding intervention will consist of a projection of future risk of co-morbidities. A visual projection model will be built using archival data available through the Singapore Diabetes Registry. The projection model will use the current profile of the participant to calculate a risk profile for the participant's potential complications and co-morbidities, which will be presented as a pie chart. The tool will also present alternative scenarios to the participant and visualize how the likelihood of complications or co-morbidities would decrease or increases if his/her habits changed. This will provide the motivational aspect of the intervention.
  This intervention takes place during Cycle 2 (second 14 weeks).
  Arms: Fast-forwarding; Fast-forwarding with weekly nudge in Cycle 1; Fast-forwarding with weekly nudge in Cycle 2; Full intervention
Behavioral: Goal-Setting plus Weekly Nudge in Cycle 2 — The procedure for goal-setting will start with the participant receiving a list of possible goals. The moderator will go through the list with the participant to identify which goals the participant is comfortable with and could reasonably achieve, and to tick off those goals that the participant has already achieved. The participants will choose their own goals. In each subsequent week, the moderator will check-in with the participant and tick off the goal(s) that have been achieved.
  Chat groups of 10-15 people will be formed to administer the weekly nudge. The participants will be encouraged to introduce themselves and to interact with each other during each the chat session. Every week for the following 14 weeks, the moderator will post diabetes-related content on the WhatsApp chat group and introduce topics of interest according to a planned schedule.
  This intervention takes place during Cycle 2 (second 14 weeks).
  Arms: Fast-forwarding with weekly nudge in Cycle 2; Full intervention; Weekly nudge; Weekly nudge in Cycle 2

SUMMARY:
Effective control of diabetes requires patients to change their daily behaviour. The investigators propose an intervention programme for behavioural change with two components, targeting motivation and implementation. The motivation component raises the salience of probable patient-specific detrimental future outcomes by 'fast-forwarding' awareness of these outcomes to the present. The implementation component helps patients to set goals and to act based on weekly tips. A factorial design will be used to establish the necessity and sufficiency of the two components on changing mind and guiding behaviour to improve blood glucose level. Individual-level measures of psychological, physical and medical conditions will be shown to drive the heterogenous responses to the two components. Intervention is expanded into two cycles with crossover design to demonstrate how the individual-level measures drive the wear-off, built-up and persistence of the two components. The results of this two-component programme will serve as a basis for systematic synthesis of component-level effectiveness in behavioural intervention research.

DETAILED DESCRIPTION:
This behavioural-change-intervention programme will be an online 'single-centre' outpatient randomized controlled trial (RCT) with ten study arms. It will be a two-component intervention consisting of a motivation component of fast-forwarding and an implementation component of goal-setting and weekly nudges. The field intervention will be structured into a two-cycle four-treatment crossover design with four treatment conditions in the first cycle and crossing-over into eight treatment conditions (including one control condition) in the second cycle. In addition to the control group in the study, a group of patients from the Singapore Health Services (SingHealth) Diabetes Registry dataset will be identified using propensity scoring to serve as a 'match-pair' for each study participant. The electronic medical record of this match-pair will provide an additional benchmark of biological measure in addition to that provided by the control group.

The field study will run for 34 weeks, in two cycles of 14 weeks each, with a 2-week transition period between the two cycles. There will also be a 2-week baseline period in which baseline measurements will be taken before the first cycle begins and a 2-week debriefing period where the final measurement will be taken after the end of the second cycle. Measurements will be taken three times: once before Cycle 1 (as the baseline), once between Cycles 1 and 2, and once at the end of Cycle 2. Participants who are assigned to the motivation component of fast-forwarding will receive fast-forwarding immediately after the measurement session and before the cycle. The participants who are randomly assigned to treatment conditions, including the implementation component, will receive a weekly nudge programme with each 14-week cycle. All participants will have access to the resources used to generate the 14-week cycles.

The investigators will measure the following: (i) physiological and medical information related to the progression of diabetes; (ii) diet quality and exercise level; (iii) psychological reactions towards diabetes management; (iv) behavioural change readiness and commitment; and (v) lifestyle (smoking, alcohol consumption, and sleep quality).

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-70
* Has type 2 diabetes
* Comfortable communicating English
* Uses smartphone app WhatsApp

Exclusion Criteria:

* Participants with diagnoses of mental health illnesses
* Participants who are unable to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c after Cycle 1 | Measured between Weeks 17-18
  Results from HbA1c test
HbA1c after Cycle 2 | Measured between Weeks 33-34
  Results from HbA1c test

SECONDARY OUTCOMES:
Diet quality after Cycle 1 | Measured between Weeks 17-18
  Diet quality will be measured using the well-validated Food Frequency Questionnaire
Diet quality after Cycle 2 | Measured between Weeks 33-34
  Diet quality will be measured using the well-validated Food Frequency Questionnaire
Exercise levels after Cycle 1 | Measured between Weeks 17-18
  Exercise level will be assessed based on the Global Physical Activity Questionnaire (GPAQ) developed by the World Health Organization in 2002 for chronic disease risk-factor surveillance
Exercise levels after Cycle 2 | Measured between Weeks 33-34
  Exercise level will be assessed based on the Global Physical Activity Questionnaire (GPAQ) developed by the World Health Organization in 2002 for chronic disease risk-factor surveillance
Attitudes towards diabetes management after Cycle 1 | Measured between Weeks 17-18
  The participants' psychological reactions towards diabetes treatment will be captured using three main groups of questionnaires. Their general attitudes towards diabetes will be measured using the Diabetes Attitude Survey developed and validated by the University of Michigan Diabetes Research and Training Center (MDRC). The investigators will measure how strongly the patients feel empowered to cope with and manage diabetes, which is a crucial outcome of DSME. Empowerment will be captured using the Diabetes Empowerment Scale (DES) developed by the MDRC. To gain insight into the psychological processes through which fast-forwarding and implementation influence health outcomes, the investigators will measure attitudes towards perceived barriers to diet adherence, exercise, and monitoring, using the respective subscales of the Diabetes Care Profile developed by MDTC
Attitudes towards diabetes management after Cycle 2 | Measured between Weeks 33-34
  The participants' psychological reactions towards diabetes treatment will be captured using three main groups of questionnaires. Their general attitudes towards diabetes will be measured using the Diabetes Attitude Survey developed and validated by the University of Michigan Diabetes Research and Training Center (MDRC). The investigators will measure how strongly the patients feel empowered to cope with and manage diabetes, which is a crucial outcome of DSME. Empowerment will be captured using the Diabetes Empowerment Scale (DES) developed by the MDRC. To gain insight into the psychological processes through which fast-forwarding and implementation influence health outcomes, the investigators will measure attitudes towards perceived barriers to diet adherence, exercise, and monitoring, using the respective subscales of the Diabetes Care Profile developed by MDTC
Readiness for behavioral change after Cycle 1 | Measured between Weeks 17-18
  To assess readiness for behavioural change, the investigators will ask the participants to indicate their commitment to make changes to their diet and physical activity. Specifically, the investigators will ask them to name a food that they have been told to eat less of, and to indicate how many times they are willing to cut back on the food. Similarly, the investigators will ask the participants to indicate how much time per week they are willing to exercise to avoid future complications arising from their diabetes
Readiness for behavioral change after Cycle 2 | Measured between Weeks 33-34
  To assess readiness for behavioural change, the investigators will ask the participants to indicate their commitment to make changes to their diet and physical activity. Specifically, the investigators will ask them to name a food that they have been told to eat less of, and to indicate how many times they are willing to cut back on the food. Similarly, the investigators will ask the participants to indicate how much time per week they are willing to exercise to avoid future complications arising from their diabetes
Smoking status after Cycle 1 | Measured between Weeks 17-18
  Self-reported smoking status
Smoking status after Cycle 2 | Measured between Weeks 33-34
  Self-reported smoking status
Level of alcohol consumption after Cycle 1 | Measured between Weeks 17-18
  Self-reported frequency of alcohol consumption
Level of alcohol consumption after Cycle 2 | Measured between Weeks 33-34
  Self-reported frequency of alcohol consumption
Sleep quality after Cycle 1 | Measured between Weeks 17-18
  Self-reported quality of sleep
Sleep quality after Cycle 2 | Measured between Weeks 33-34
  Self-reported quality of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Investigators will not be storing or sharing any personal identifiers. All individual level data will be anonymized, and only anonymized data will be shared with other researchers, upon request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The supporting information will be made available upon publication in the supporting documentation.
Access Criteria: It will be made available in the supporting documentation.